CLINICAL TRIAL: NCT06068699
Title: Informational Postcards to Improve Remote Monitoring Among Veterans With Pacemakers and Implantable Cardioverter-Defibrillators
Brief Title: Postcards to Improve Remote Monitoring Adherence Among Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Sanket Dhruva, MD, MHS, Staff Physician, San Francisco VA Health Care System
Organization: San Francisco VA Health Care System (U.S. Federal Agency)
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Health Services Research
Other Study IDs: VANCDSP QUERI Postcards
Record Dates: First submitted 2023-09-21; First posted 2023-10-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-09

CONDITIONS: ICD; Pacemaker DDD; Adherence, Patient
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Intervention Model Description: This was a stepped-wedge randomized controlled trial with two waves. In wave 1, Veterans who had sent at least 1 transmission within the past 2 years but had become non-adherent were randomly assigned to receive a postcard or no postcard. Those receiving postcards were randomized to 1 of 2 messages: 1) a "warning" postcard describing risks of non-adherence or 2) an "encouraging" postcard describing benefits of adherence. In wave 2, Veterans who had either not received a postcard in wave 1 or had since become non-adherent were mailed a postcard (again, randomized to 1 of 2 messages). Patients who did not send a RM transmission within 1 month were mailed a second, identical postcard.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Postcards (Experimental): Participants who received a postcard.
  Interventions: Other: Postcard
- Controls (No Intervention): Participants did not receive a postcard (usual care).

INTERVENTIONS:
Other: Postcard — Participants received a postcard asking them to address non-adherence to remote monitoring.
  Arms: Postcards

SUMMARY:
We tested the effect of informational postcards on improving remote monitoring adherence among Veterans with pacemakers and implantable cardioverter-defibrillators in a stepped-wedge randomized controlled trial.

DETAILED DESCRIPTION:
Objective: To test the effect of informational postcards on remote monitoring adherence among Veterans with pacemakers and implantable cardioverter-defibrillators (ICDs).

Design/Patients: Stepped-wedge randomized controlled trial among Veterans with pacemakers and ICDs.

Intervention: In wave 1, Veterans who had sent at least 1 transmission within the past 2 years but had become non-adherent were randomly assigned to receive a postcard or no postcard. Those receiving postcards were randomized to 1 of 2 messages: 1) a "warning" postcard describing risks of non-adherence or 2) an "encouraging" postcard describing benefits of adherence. In wave 2, Veterans who had either not received a postcard in wave 1 or had since become non-adherent were mailed a postcard (again, randomized to 1 of 2 messages). Patients who did not send a remote monitoring transmission within 1 month were mailed a second, identical postcard.

Main Measures: Proportion of patients who sent a transmission within 70 days.

ELIGIBILITY:
Inclusion Criteria:

* Veteran patients with wireless RM-capable pacemakers and ICDs followed by the VA National Cardiac Device Surveillance Program (VANCDSP)
* Sent at least 1 remote transmission within the past 2 years but had become non-adherent (defined as missing their last scheduled transmission by at least 10 days)

Exclusion Criteria:

* Veteran patients without a wireless RM-capable device
* Had not sent a remote transmission in the past 2 years

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6351 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Remote monitoring transmission | 70 days
  Proportion of patients who sent a transmission within 70 days

SECONDARY OUTCOMES:
Transmission after first postcard | 70 days
  Proportion of patients who sent a transmission after the first postcard

CONTACTS AND LOCATIONS:
Locations (1):
- San Francisco VA Medical Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No